CLINICAL TRIAL: NCT07282951
Title: Strong Evidence: Randomized Digitally Delivered Fall-Prevention Exercise Trial in Older Adults
Brief Title: Strong Evidence: Digitally Delivered Exercise in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Sanford Burnham Prebys (Other)
Responsible Party: Principal Investigator, Ryan Moran, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 812960
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Fall Prevention; Fall Prevention in Healthy Aging
Keywords: Fall Prevention; Digital Exercise; Digital; Group Exercise; Exercise; Older Adults; Fracture prevention; Balance; Strength; Posture
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: As such individuals will be randomized by cohort into either
  * Group A: who will start their 12-week exercise program with the Intensive Intervention within 4 weeks of baseline measurement. For those who qualify (see below) this will be followed by a 12-week maintenance program. This group will finish the program with 12 weeks life as usual.
  * Broup B: who willl have a 12 week lead in period of life as usual. They will then begin their 12-week intensive intervention. Those who qualify, this will be followed by a 12-week maintenance program.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention: Group A (Experimental): • Group A: who will start their 12-week exercise program with the Intensive Intervention within 4 weeks of baseline measurement. For those who qualify (see below) this will be followed by a 12-week maintenance program. This group will finish the program with 12 weeks life as usual.
  Interventions: Behavioral: Digitally Delivered Exercise
- Delayed Intervention: Group B (Experimental): • Broup B: who willl have a 12 week lead in period of life as usual. They will then begin their 12-week intensive intervention. Those who qualify, this will be followed by a 12-week maintenance program.
  Interventions: Behavioral: Digitally Delivered Exercise

INTERVENTIONS:
Behavioral: Digitally Delivered Exercise — Our fall- risk reduction program, Strong Foundations, was designed to be delivered digitally, and while there are many such programs currently available on the Internet, especially in the time of COVID-19, the novel feature of this program is the delivery of semi-individualized instruction in real time within a small group setting.
  The program was designed with physician input and by exercise physiologists and a Doctor of Physical Therapy candidate, all with extensive training in both group and individualized exercise for geriatric populations.
  Strong Foundations is a 12 week iterative curricular program with three core components: postural alignment and control, balance and mobility, and muscular strength and power. All the exercises offered over the course of the intervention are appropriate for the target population and are standardized so all participants receive the same basic instruction, but level of difficulty is scaled to participant capability.
  Other Names: Strong Foundations

SUMMARY:
The investigators have successfully completed a pilot project focused on feasibility and user acceptability of a digitally delivered program for fall prevention in older adults. It was well received among a population of lower and moderate risk individuals. The investigators propose to extend this research by repeating the training program with the inclusion of a wait list control group.

Group A (immediate intervention) will start their initial 12 week exercise program (Intensive Exercise) within 4 weeks of baseline (BL) measurement (as a cohort). This will be followed by an optional additional 12 week exercise program (Maintenance Exercise 2) that participants who complete at least 10 of the Exercise 1 classes will be invited to join. This will be followed by a 12 week wash out period. Measurements will occur each 12 weeks (BL, 12 week post randomization, 24 week post randomization, 36 week post randomization)

Group B (waitlist control) will start with a 12 week life as normal period that is concurrent with Group A's intensive Exercise. They will start Intensive Exercise when Group A is doing Maintenance exercise. They will be invited to Maintenance Exercise while Group A is doing washout. They will not have a washout period. Measurements will occur at the same period(s) as Group A (i.e. all participants measured during the same time period).

The intervention will be identical to what was offered in the past, and measurements will be very similar (removing those that did not show change with intervention or were deemed too difficult for participants).

DETAILED DESCRIPTION:
While fall risk is multifactorial, identification of risk factors and referral to/participation in appropriate fall-risk reduction programs are established as an effective, evidenced-based approach to reduce fall-risk. Specifically, targeted strength and balance exercise have consistently been shown to improve fall risk, and accordingly, the Centers for Disease Control and Prevention (CDC) has outlined an evidenced-based clinical approach to identify those at risk for falls to help assess known risk factors and to refer for community-based fall-prevention programs. This toolkit, however, has been slow to penetrate in routine clinical practice, as barriers reported by physicians to implementing comprehensive falls-prevention screening are time constraints, poor reimbursement for falls screening, and that existing toolkit utilization does not easily fit into a Medicare wellness visit. Because of this, only approximately one-third of older adults report being asked about fall-risk, and similarly only around a third of those who fall report discussing this with their healthcare provider. Compounding this, COVID-19 has created uncertainty in accessing community resources, increased sedentary behavior, isolation and subsequent fall risk. This is especially disconcerting as a single fall predicts recurrent falls with between 10% and 44% of elderly patients with a history of falls sustaining additional falls within five years.

COVID-19 has confounded social isolation in older adults, especially those in congregate settings. Appropriate technology/technologic driven approaches has promise (but limitations) to mitigate some aspects of loneliness/isolation in this population. Digitally delivered programs are an opportunity that help balance risks and benefits during times of social distancing, improve dissemination, and possibly improve objective measures of function. Therefore, approaches to improve access to fall-risk reduction exercise, including balance and strength training opportunities is imperatively important, and growing data suggests digitally formatted delivery may be feasible.

This project also offers the potential to expand our knowledge regarding successful aging using the basic sciences. Specifically, autophagy is the process by which the body packages and recycles damaged proteins and organelles making it essential for maintaining proteostasis and cellular quality control. Autophagy is a dynamic, multi-step process, and static measurements (e.g., protein levels) are insufficient to distinguish increased flux from impaired degradation. Recently, assays of autophagy flux in peripheral blood mononuclear cells (PBMCs) have been developed, enabling minimally invasive, reproducible measurement of this process in human cohorts, but there has currently been limited application to human models. Thus, this project creates a unique opportunity to begin linking autophagy biology with functional outcomes in older adults. Even more meaningfully, autophagy flux in PBMCs has not yet been assessed after any form of exercise, despite the known impact of exercise on functional outcomes and resilience. Establishing PBMC autophagy flux as a biomarker of resilience in this context would address a major translational gap, bridging basic mechanisms of aging biology with functional outcomes of intervention and help guide strategies to maintain health and independence in older adults.

Fall Prevention Program: Our fall- risk reduction program, Strong Foundations, was designed to be delivered digitally, and while there are many such programs currently available on the internet, especially in the time of COVID-19, the novel feature of this program is the delivery of semi-individualized instruction in real time within a small group setting. This is accomplished largely by use of the 'breakout room' feature on the Zoom platform, where 2-3 trained intern instructors correct form while the lead instructor teaches the larger group. The program was designed with physician input and by exercise physiologists and a Doctor of Physical Therapy candidate, all with extensive training in both group and individualized exercise for geriatric populations. Strong Foundations is a 12 week iterative curricular program with three core components: postural alignment and control, balance and mobility, and muscular strength and power. All the exercises offered over the course of the intervention are appropriate for the target population and are standardized so all participants receive the same basic instruction, but level of difficulty is scaled to participant experience, capability, and musculoskeletal limitations.

While many exercise interventions for fall prevention have been validated in different populations, our program is designed with the community in mind and with a novel platform to improve dissemination/availability across many populations.

ELIGIBILITY:
Inclusion Criteria:

* Has the capacity to provide informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 60 or older, ambulatory, including with the use of a cane or walker, and able to read and speak English.
* Access to internet/computer and Zoom-interface / broadband with a device with a minimum screen size of 7 inches (i.e. tablet or larger).
* Completion of the Stopping Elderly Accidents, Deaths & Injuries (STEADI) Stay Independent Risk for Falling Questionnaire (uploaded as Supporting materials). NOTE: A score of 7 or greater will make a participant ineligible for this study (see below).

Exclusion Criteria:

* Individuals who are wheel-chair bound
* Score 7 or more on the STEADI Risk for Falling questionnaire.
* Individuals who have non removable (i.e. implanted) electrically driven medical implants (pacemakers, cochlear implants, etc)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
30 second chair stand | Baseline, 12 weeks, 24 weeks, 36 weeks
  The 30-Second Chair Stand is intended to evaluate lower body and hip flexor strength and short endurance. This assessment is easy and quick to administer, and has been shown to predict falls with cut-offs that are age and gender adjusted. Individuals are instructed to sit in in an arm-less chair of approximately 17 inch seat-height, cross their arms across the chest, keep their feet flat on the floor and back straight, and sequentially rise and sit as many times as possible within a 30-second time frame

SECONDARY OUTCOMES:
Grip Strength | Baseline, 12 weeks, 24 weeks, 36 weeks
  Hand grip strength will be measured in both hands using an adjustable grip strength dynamometer that quantifies force in kilograms (BL5001 Hydraulic Hand Dynamometer). The grip bar of the instrument will be adjusted so the second joint of the fingers first snugly under the handle and the hand position will be recorded (1-5). The dynamometer will be set to zero and the participant will be given a chance to familiarize themselves with the measurement by giving a submaximal effort on both hands to feel how the instrument will react. For the assessment, the participant will stand and hold the dynamometer in their hand with their arm down at their side. The participant will be instructed to take a deep breath in, and squeeze as hard as possible as they exhale. The measurement will be repeated twice on each hand, alternating between each side, and the highest score for each hand will be recorded to the nearest kilogram.
Occipital to Wall Distance | BL, 12 weeks, 24 weeks, 36 weeks
  b) Occipital to Wall Distance (OWD) will be measured with participants standing with their feet together and their heels and buttocks touching the wall while they look forward (or as close to the wall as possible. The distance from the wall to their occiput (back of the head) will be measured to the nearest 0.1 cm. Measurements will be taken twice, with a third measurement gathered in the event that there is greater than 0.3 cm difference between the first two measures. An average of the closest two measurements will be used for analysis. Pictures will be captured via Zoom to collect this measure.
Short Physical Performance Battery (SPPB) | Baseline, 12 weeks, 24 weeks, 36 weeks
  The Short Physical Performance Battery (SPPB) measures gait speed, leg strength (via chair stand time) and the three stage balance assessment recommended by the CDC for assessing fall risk. This composite measure includes evaluating side-by-side, semi-tandem, and tandem position, time to walk 4 meters , and time to rise from a chair and return seated five times.
  Each of these (sub)measures are categorically scored from 0-4 with a composite score from 0-12 and higher numbers being indicative of superior function.
The Timed Up and Go (TUG) | Baseline, 12 weeks, 24 weeks, 36 weeks
  The Timed up and Go (TUG) is an easy to administer office-based assessment in which a person rises from a seated position without using their arms, walks three meters (approximately 10 feet), turns around, returns to the chair, and sits down while being timed. The TUG has been found to be reliable with good inter-rater and intra-rater reproducibility, and is a good predictor of frailty. While there is some disagreement regarding its role in falls-prediction, the CDC suggests a cutoff time of 12 seconds to discriminate fall risk. This will be performed twice and the better of the two scores recorded.
  Faster speeds (i.e. shorter times) are indicative of superior function
Body Muscle | Baseline, 12 weeks, 24 weeks, 36 weeks
  d) Body Composition will be measured by bioelectrical impedance analysis (BIA) using a Tanita DC-430U Dual Frequency Total Body Composition Analyzer (device manual included as attachment). This machine looks like a doctor's scale, but it also measures body composition using a weak constant current source with a high frequency current (6.25kHz, 50kHz, 90μA), which is not a significant amount of energy. The 4 electrodes are positioned so that electric current is supplied from the electrodes on the tips of the toes of both feet, and voltage is measured on the heel of both feet.
  Values are provided for absolute mass of lean tissue (muscle), fat tissue, and bone and percentage of body fat is derived. In general, larger amounts of lean tissue, and lower percentage body fat are indicative of better health and function.
Autophagy Flux | Baseline, 12 weeks, 24 weeks, 36 weeks
  e) Autophagy Flux will be measured in freshly isolated human peripheral blood mononuclear cells (PBMCs). A trained phlebotomist will draw 9 mL of fasting blood into Vacuette lithium heparin tubes using standard venipuncture. Freshly-drawn whole blood will be treated with the late-stage autophagy inhibitor chloroquine, after which peripheral blood mononuclear cells (PBMCs) will be isolated, lysed, and analyzed by Western blot.
  Autophagy flux is a continuous biomarker without established clinical thresholds. Interpretation focuses on within-subject change over time and correlations with functional outcomes rather than absolute values.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Kumstra, PhD, Principal Investigator — Sanford Burnham Prebys; Ryan Moran, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are currently undecided about sharing individual-level participant data (IPD) from this exercise intervention. It is likely that deidentified data regarding strength, balance, and autophagy flux at all timepoints will be shared.
  In the event that materials are shared the investigators will provide deidentified datasets based upon a application to use data to replicate or publish which includes a clear research plan and use for the data.
  Provided data will be deidentified, and data that is not required for the specific research question/plan will not be included.

REFERENCES:
- [Background] Bansal S, Katzman WB, Giangregorio LM. Exercise for improving age-related hyperkyphotic posture: a systematic review. Arch Phys Med Rehabil. 2014 Jan;95(1):129-40. doi: 10.1016/j.apmr.2013.06.022. Epub 2013 Jul 9. PMID 23850611
- [Background] Wing D, Nichols JF, Barkai HS, Culbert O, Moreno D, Higgins M, O'Brien A, Perez M, Davey H, Moran R. Building Strong Foundations: Nonrandomized Interventional Study of a Novel, Digitally Delivered Fall Prevention Program for Older Adults. JMIR Aging. 2025 Feb 26;8:e68957. doi: 10.2196/68957. PMID 40009847
- [Background] Jacobson CL, Foster LC, Arul H, Rees A, Stafford RS. A Digital Health Fall Prevention Program for Older Adults: Feasibility Study. JMIR Form Res. 2021 Dec 23;5(12):e30558. doi: 10.2196/30558. PMID 34837492
- [Background] Gill TM. Assessment of function and disability in longitudinal studies. J Am Geriatr Soc. 2010 Oct;58 Suppl 2(Suppl 2):S308-12. doi: 10.1111/j.1532-5415.2010.02914.x. PMID 21029059
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Sarmiento K, Lee R. STEADI: CDC's approach to make older adult fall prevention part of every primary care practice. J Safety Res. 2017 Dec;63:105-109. doi: 10.1016/j.jsr.2017.08.003. Epub 2017 Sep 4. PMID 29203005
- [Background] Stevens JA, Phelan EA. Development of STEADI: a fall prevention resource for health care providers. Health Promot Pract. 2013 Sep;14(5):706-14. doi: 10.1177/1524839912463576. Epub 2012 Nov 16. PMID 23159993

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT07282951/Prot_SAP_000.pdf